CLINICAL TRIAL: NCT04796558
Title: Validation of Arterio Venous Access Stage Classification by Using Machine Learning in Prediction of Vascular Access Creation and Uninterrupted Use of the Vascular Access for Dialysis
Brief Title: Validation of Arterio Venous Access Stage (AVAS) Classification
Acronym: VAVASC
Status: Active, not recruiting | Type: Observational
Sponsor: Vascular surgery, University hospital Královské Vinohrady, Prague (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 532021
Record Dates: First submitted 2021-03-05; First posted 2021-03-15 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Arteriovenous Graft; Arteriovenous Fistula; Dialysis Access Malfunction; Kidney Failure; Dialysis Related Complication
Keywords: Arterio venous access; Dialysis; AVAS; Predictive modelling; Machine learning; VAVASC; Multicentre; Observational; Prospective
MeSH Terms: conditions — Arteriovenous Fistula; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AVAS Classification — Validation of AVAS classification

SUMMARY:
VAVASC trial is an observational multicentre study. The aim of this trial is to validate AVAS (arteriovenous vascular access stage) classification. The classification is used for determining which type of access is the most suitable for the patient on the basis of the patient´s vascular anatomy

The methodology of this trial is to apply AVAS classification on patients who are indicated for creation of vascular access for hemodialysis. Data on these patients (vascular anatomy status, AVAS type, and predicted type of arterio venous access, demographic data etc.) will be than statistically analysed. Patients will then undergo creation of the selected arteriovenous access. They will be observed in terms of the access functionality. The follow up will be 1 to 3 years. The second aim of this study is to evaluate the relationship between AVAS classification and uninterrupted use of the created arterio venous access.

DETAILED DESCRIPTION:
Ultrasound of upper limb vessels as a part of preoperative assessment of patients referred for arteriovenous access placement has been recommended repeatedly in several studies and guidelines. Each patient needing arterio-venous access (AVA) is unique and has different possibilities for fistula creation that depend on many factors as well the anatomical condition of inflow arteries and outflow veins, the so-called 'arteriovenous access map'. In 2020 we created, published and retrospectively evaluated the inter-rater reliability of the AVAS classification, which is a simplified way of sharing the information about suitability for access creation depending on vascular anatomy (doi: 10.1093/ckj/sfaa189).

However, before routine use of the AVAS classification system in clinical practise it requires prospective validation and comparison with other clinical factors. Finally, whether the AVAS classification can be used for the prediction of vascular access function as defined by uninterrupted use of vascular access for dialysis without need for any access intervention/procedures (SONG-HD, doi: 10.1053/j.ajkd.2017.12.003) remains to be tested.

This project has two main parts:

1. Validation of AVAS classification with and without combination with other factors using a predictive statistical model

   .
2. Validation of AVAS classification in terms of prediction of uninterrupted use of successfully created vascular access for dialysis.

The data will be collected prospectively. Both parts of the project will be taking place simultaneously.

Data will be collected prospectively (Belfast City Hospital, UK, University hospital Královské Vinohrady Prague CZ). Other centres around the world will be asked for cooperation (announcement will be posted via Twitter, ResearchGate, LinkedIn, Facebook and Kidney Academy) in January 2021. The data collected will be the parameters of the vessels on the upper limb, in order to be able to evaluate AVAS (VAVASC FORM). Along with anatomical dispositions of the patients, other parameters will be collected.

Obligatory parameters (parameters A):

Side of the arm (Left / Right) Dominant hand (Left / Right) Allen's test (Positive / Negative) (A negative Allen's test is demonstration of a complete palmar arch and intact collateral blood flow to the hand) Sex(M / F) Age, Height, Weight, BMI, Diabetes (Yes / No) Central venous line previous or current (Yes / No) Side of the central venous line if place (Left / Right)

Non-obligatory parameters (parameters B):

Smoking history (Yes / No) Hypertension (Yes / No) Heart failure (Yes / No) Ischemic heart disease (Yes / No) Cancer (previous or current) (Yes / No)

In order to evaluate uninterrupted use of the vascular access for dialysis (part 2 of the study), we will follow the patients and do a time to event analysis of the arteriovenous accesses for one year after creation or up until the first intervention for maintaining patency has been performed. If the patient dies during follow up the date of death should be recorded. The data for this part will be collected prospectively (Belfast City Hospital, UK, University hospital Královské Vinohrady Prague, CZ and other centres).

Predictive models will be used for validation of AVAS classification. The data will be registered via electronic database and analysed by Waldauf, P. and O'Neill, S.

ELIGIBILITY:
Inclusion Criteria:

* patients indicated for creation of arterio venous access for dialysis

Exclusion Criteria:

* patients who disagree to participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - patients with kidney insufficiency who are indicated for creation of arterio venouss access for dialysis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Arterio Venous Access Stage (AVAS) evaluation | Baseline - recruiting (Year 1) - physical examination, data collection and evaluation of Arterio Venous Access Stage (AVAS)
  What type of the Arterio Venous Access Stage (AVAS classification) the patient has based on his/her vascular anatomy of upper limbs
Arterio Venous Access type predicted | Baseline - recruiting (Year 1) - physical examination, data collection and evaluation of Arterio Venous Access Stage (AVAS) and predicting a type of arterio venous access
  What type of the Arterio Venous Access is predicted based on AVAS and other clinical factors
Final Arterio Venous Access | Follow up (up to 1-2 years) what type of arterio venous access was eventually created
  What type of the arterio venous access was eventually created (in corelation with AVAS evaluation and the predicted arteriovenous access type)
Functionality of the arterio venous access | Year 2-3 - follow up, collection the data about the functionality (uninterrupted use) of the arterio venous access and evaluation of the relation between AVAS and the functionality of the arterio venous access
  Uninterrupted use of the created arterio venous access

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular surgery, University hospital Královské Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lawrie K, Waldauf P, Balaz P, Bortel R, Lacerda R, Aitken E, Letachowicz K, D'Oria M, Di Maso V, Stasko P, Gomes A, Fontainhas J, Pekar M, Srdelic A; VAVASC Study Group; O'Neill S. Machine learning validation of the AVAS classification compared to ultrasound mapping in a multicentre study. Sci Rep. 2025 Jan 20;15(1):2538. doi: 10.1038/s41598-025-86456-3. PMID 39833325
- [Derived] Katerina L, Stephen O, Petr W, Peter B. VAVASC study: Clinical trial protocol. J Vasc Access. 2023 Jul;24(4):792-797. doi: 10.1177/11297298211042677. Epub 2021 Sep 2. PMID 34472988
- See also: Related Info — https://www.vavasc.com/

DOCUMENTS (1):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT04796558/Prot_000.pdf